CLINICAL TRIAL: NCT05248204
Title: Prospective, Randomized, Split-mouth Study Evaluating Clinical Performance of 3M™ Scotchbond™ Universal Plus Adhesive Compared to 3M Scotchbond Universal Adhesive for Posterior Class I & II Restorations With 3M Filtek™ Universal Restorative
Brief Title: Scotchbond Universal Plus Compared to Scotchbond Universal for Posterior Class I & II Restorations With Filtek Universal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EM-11-050069
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Cavities of Teeth; Dental Decay
Keywords: dental materials; dental adhesives; dental fillings; dental cavities; Scotchbond Universal Plus; Scotchbond Universal; Filtek Universal Restorative
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, open-label, assessor-blinded, split-mouth, single-center post-market clinical follow-up study.
Who Masked: Outcomes Assessor
Masking Description: All assessments will be performed by two dental examiners that are independent of the dentist that placed the restorations and are blinded to the treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Scotchbond Universal Plus Treatment (Experimental): Study tooth with posterior Class I or Class II carious lesion randomized to undergo restoration using Scotchbond Universal Plus (SBU+) Adhesive (Treatment).
  Interventions: Device: Scotchbond™ Universal Plus Adhesive
- Scotchbond Universal Comparator (Active Comparator): Study tooth with posterior Class I or Class II carious lesion randomized to undergo restoration using the predicate device, Scotchbond Universal (SBU) Adhesive (Control).
  Interventions: Device: Scotchbond™ Universal Adhesive

INTERVENTIONS:
Device: Scotchbond™ Universal Plus Adhesive — Eligible tooth with Class I or Class II carious lesion randomized to the SBU+ treatment group will undergo restoration with Scotchbond™ Universal Plus Adhesive using self-etch mode and Filtek Universal Restorative
  Arms: Scotchbond Universal Plus Treatment
Device: Scotchbond™ Universal Adhesive — Eligible tooth with Class I or Class II carious lesion randomized to the SBU control group will undergo restoration with Scotchbond™ Universal Adhesive using self-etch mode and Filtek Universal Restorative
  Arms: Scotchbond Universal Comparator

SUMMARY:
This research study is looking at a new bond-promoting substance (a dental adhesive called 3M™ Scotchbond™ Universal Plus Adhesive) used between the tooth and dental restoration (filling). This is a randomized, split-mouth study designed to evaluate whether Scotchbond™ Universal Plus Adhesive (SBU+) is as effective at bonding dental fillings as Scotchbond™ Universal Adhesive (SBU) for preparation of posterior Class I and Class II restorations in adult patients. Participants must have at least two (2) back teeth that need a filling either on the chewing surface alone (Class I) and/or on the chewing surface and between your teeth (Class II). One tooth will be restored using SBU+ and the other tooth will be restored using SBU adhesive, both filled using Filtek™ Universal Restorative as the filling material.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, open-label, assessor-blinded, split-mouth, single-center post-market clinical follow-up study. The study is designed to compare the clinical efficacy of Scotchbond™ Universal Plus Adhesive with Scotchbond™ Universal Adhesive when used in self-etch mode for preparation of posterior Class I and Class II restorations using Filtek™ Universal Restorative material in adult patients.

Selected endpoints are based partly on the FDI World Dental Federation criteria. Subjects who meet all inclusion and none of the exclusion criteria and who have provided informed consent will be eligible for enrollment and must be treated within 21 days of screening. Either two pre-molars or two molars from each Subject will be randomized in a 1:1 ratio such that one of the teeth will be randomized to undergo restoration using SBU+ Adhesive (Treatment), and the other tooth will undergo restoration using SBU Adhesive (Control). Both study teeth will be restored using Filtek™ Universal Restorative material as the filling material. Individual subject participation is expected to last 2 years (± 45 days) with scheduled study visits at screening, day of restoration/baseline, and follow-up visits at 6 months (± 14 days), 1 year (± 30 days), and 2 years (± 45 days) after restoration. The entire duration of the study is expected to last approximately 3 years, with individual Subject participation expected to last up to 2 years (± 45 days).

To help minimize or avoid bias in the study, randomization of study teeth will occur after teeth preparation but before the initial application of any adhesive. All assessments will be performed by two dental examiners that are independent of the dentist that placed the restorations and are blinded to the treatment arms. All examiners will be trained and calibrated for the scoring criteria before any Subject assessment occurs, and examiners will be retrained and recalibrated if any new evaluator is added to the list of assessors. After the second examiner has completed their assessments, then the examiners will compare their evaluations and a consensus will be reached for each of the scoring criteria at each visit. A consensus will be reached before the Subject leaves the visit, and the consensus assessments will be entered into the Case Report Form (CRF).

ELIGIBILITY:
Inclusion Criteria:

1. The Subject is between the ages of 18 and 70 years old at time of consent.
2. The Subject requires at least two direct composite restorations for posterior Class I or Class II carious lesions in vital teeth that are asymptomatic and with minimal mobility (< 1 mm in the buccolingual direction).
3. Study teeth have a minimum buccolingual diameter of the occlusal surface that is at least 1/3 of the distance between the buccal and lingual cusps
4. Teeth selected for Class II restorations need to have an adjacent tooth in a position that will allow for a contact relationship to be established.
5. The Subject is able and willing to sign Informed Consent Form in English without assistance.
6. The Subject is able and willing to be available for all scheduled study visits.
7. The Subject is in good general health (ie, meets American Society of Anesthesiologists (ASA) Level I or ASA Level II classification criteria).
8. The selected teeth need to have occlusal contact with an antagonistic natural tooth.
9. The Subject has existing radiographic images of the study teeth of current and acceptable diagnostic quality obtained within the previous 12 months.

Exclusion Criteria:

1. The Subject has a history of adverse reaction to any materials used in this study.
2. The Subject is pregnant or breast feeding at the time of screening.
3. The Subject has fewer than 20 teeth.
4. The Subject is taking part in or planned to be enrolled in an evaluation of other restorative materials at any time during the study.
5. The Subject has advanced periodontal disease (ie, Grace & Smales Mobility Index grade ≥ 2) that involve the study teeth.
6. The Subject had orthodontic appliance treatment within the previous 3 months.
7. The Subject has pronounced enamel wear facets, indicating severe, on-going bruxism.
8. The Subject has severe xerostomia.
9. The study tooth has a history of or existing, prolonged tooth hypersensitivity.
10. The study tooth is an abutment for fixed or removable prostheses.
11. The study tooth has a fracture or is visibly cracked such that it may impact the longevity of the tooth.
12. The carious lesion is stage RC5 or RC6 of the ICDAS radiographic scoring system.
13. The Subject is unable to understand study procedures or provide consent in English.
14. The Subject is an employee or student of the study investigator(s).

Intraoperative Exclusion Criteria:

1) The Subject has pulp exposure of either study tooth during the restoration procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Perdigao, DMD, MS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota School of Dentristry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Perdigao J, Dutra-Correa M, Anauate-Netto C, Castilhos N, Carmo AR, Lewgoy HR, Amore R, Cordeiro HJ. Two-year clinical evaluation of self-etching adhesives in posterior restorations. J Adhes Dent. 2009 Apr;11(2):149-59. PMID 19492717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient population was selected from current patients under clinical treatment at the University of Minnesota Dental School. Patients were between the ages of 18 and 70 years old at time of consent, of either sex, and of any ethnic background. Eligible patients needed to have at least two direct composite restorations for posterior (premolars or molars) Class I or Class II carious lesions in vital teeth that were asymptomatic and with minimal mobility.
Pre-assignment Details: Subjects were required to meet all inclusion and none of the exclusion criteria to be eligible for study participation. Any subject with pulp exposure of either study tooth during the restoration procedure was excluded from the study. Two Class I or Class II restorations were placed per patient. Selected study teeth were randomized in a 1:1 ratio with one tooth restored using SBU+ Adhesive (Treatment), and the other tooth restored using SBU Adhesive (Control).
Units Other Than Participants: Restorations
Period: Overall Study
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Started (A total of 51 subjects were included in the study, each with 2 Class I or Class II restorations performed. Teeth were randomized in a 1:1 ratio such that 51 teeth were restored using SBU+ Adhesive (Treatment), and 51 teeth underwent restoration using SBU Adhesive (Control) for a total of 102 restorations in the study.) | 51; 51 Restorations | 51; 51 Restorations
Completed (A total of 38 subjects completed the study. One subject had one tooth withdrawn due to non-compliance with study restrictions, for a total of 37 restorations with SBU+ and 38 restorations with SBU completing the study.) | 37; 37 Restorations | 38; 38 Restorations
Not Completed | 14; 14 Restorations | 13; 13 Restorations
Not completed — Lost to Follow-up | 13 | 13
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: 51 subjects each had 2 teeth treated in a 1:1 randomization with 1 tooth in each treatment group for a total of 102 restorations.
Units Other Than Participants: Restorations
Groups:
- Total: Total of all reporting groups
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator | Total
Number analyzed (Participants) | 51 | 51 | 51
Number analyzed (Restorations) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (12.4) | 33 (12.4) | 33 (12.4)
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0
  19 years to 64 years | 50 | 50 | 50
  >= 65 years | 1 | 1 | 1
Sex/Gender, Customized [Number; unit: Participants]
  Female | 28 | 28 | 28
  Male | 23 | 23 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 9 | 9 | 9
  Race: Black or African American | 12 | 12 | 12
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 23 | 23 | 23
  Race: Other | 3 | 3 | 3
  Race: Multiple Race | 4 | 4 | 4
  Ethnicity: Hispanic or Latino | 5 | 5 | 5
  Ethnicity: Not Hispanic or Latino | 44 | 44 | 44
  Ethnicity: Unknown or Not Reported | 2 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 51
Tooth Characteristic: Restoration Class [Count of Units; unit: Restorations] — Population: 51 subjects each had 2 teeth treated in a 1:1 randomization with 1 tooth in each treatment group for a total of 102 restorations (55 Class I restorations and 47 Class II restorations).
  Restorations
    Class I Restorations | 26 | 29 | 55
    Class II Restorations | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Retention of Restorative Material
Description: The percentage of restorations with partial or complete loss of the restoration materials
Time Frame: 24 months post-restoration
Population: 38 subjects completed the study; 1 subject in the treatment group had 1 tooth withdrawn prior to 24 months
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 38 | 38
Number analyzed (Restorations) | 37 | 38
percentage of restorations
  No loss of restorative material | 97 | 100
  Partial or complete loss of restorative material | 3 | 0

2. Primary Outcome: Fracture of Restorative Material
Description: Fractures on study teeth graded on a 0-4 grading scale with a score of 1 being Excellent/very good and a score of 4 being Unsatisfactory. Grading scale is based on modified FDI (Fédération Dentaire Internationale) World Dental Federation criteria.
Time Frame: 24 months post-restoration
Population: 38 subjects completed the study; 1 subject had 1 tooth withdrawn prior to 24 months
  Scoring categories for the fracture of restorative material are defined as follows:
  1. Excellent/very good: No fractures/cracks
  2. Good: Small hairline cracks
  3. Sufficient/Satisfactory: Two or more or larger hairline cracks and/or material chip fracture not affecting the marginal integrity or approximal contact
  4. Unsatisfactory: Material chip fractures which damage marginal quality or approximal contacts
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 38 | 38
Number analyzed (Restorations) | 37 | 38
percentage of restorations
  1. Excellent/Very Good | 97 | 100
  2. Good | 0 | 0
  3. Sufficient/Satisfactory | 3 | 0
  4. Unsatisfactory | 0 | 0

3. Primary Outcome: Marginal Adaptation
Description: Marginal adaptation of restorations graded on a scale of 1-5 with a score of 1 being Excellent/very good and a score of 5 being Poor. Grading scale is based on modified FDI World Dental Federation criteria.
Time Frame: 24 months post-restoration
Population: Scoring categories for marginal adaptation are defined as follows:
  1. Excellent/very good: No clinically detectable gap.
  2. Good: Marginal integrity deviates from the ideal but could be upgraded to ideal by polishing.
  3. Sufficient/satisfactory: Leakage/discoloration is present but limited to the marginal area.
  4. Unsatisfactory: Localized major gap that may result in exposure of dentine or base.
  5. Poor: Generalized major gap or irregularities; or the restoration is loose but in situ.
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 38 | 38
Number analyzed (Restorations) | 37 | 38
percentage of restorations
  1. Excellent/Very Good | 8 | 4
  2. Good | 92 | 94
  3. Sufficient/Satisfactory | 0 | 2
  4. Unsatisfactory | 0 | 0
  5. Poor | 0 | 0

4. Secondary Outcome: Retention of Restorative Material
Description: The percentage of restorations with partial or complete loss of the restoration materials
Time Frame: 6 months post-restoration
Population: Ten (10) of 51 subjects missed the 6-month follow-up visit.
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 41 | 41
Number analyzed (Restorations) | 41 | 41
percentage of restorations
  No loss of restorative material | 100 | 100
  Partial or complete loss of restorative material | 0 | 0

5. Secondary Outcome: Retention of Restorative Material
Description: The percentage of restorations with partial or complete loss of the restoration materials
Time Frame: 12 months post-restoration
Population: Six (6) of 51 subjects missed the 1-year follow-up visit. One (1) subject completed the 1-year follow-up visit, but outside the allowed time window and was excluded from this analysis.
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 44 | 44
Number analyzed (Restorations) | 44 | 44
percentage of restorations
  No loss of restorative material | 100 | 100
  Partial or complete loss of restorative material | 0 | 0

6. Secondary Outcome: Fracture of Restorative Material
Description: Fractures on study teeth graded on a 0-4 grading scale with a score of 1 being Excellent/very good and a score of 4 being Unsatisfactory. Grading scale is based on modified FDI World Dental Federation criteria.
Time Frame: 6 months post-restoration
Population: Ten (10) of 51 subjects missed the 6-month follow-up visit.
  Scoring categories for the fracture of restorative material are defined as follows:
  1. Excellent/very good: No fractures/cracks
  2. Good: Small hairline cracks
  3. Sufficient/Satisfactory: Two or more or larger hairline cracks and/or material chip fracture not affecting the marginal integrity or approximal contact
  4. Unsatisfactory: Material chip fractures which damage marginal quality or approximal contacts
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 41 | 41
Number analyzed (Restorations) | 41 | 41
percentage of restorations
  1. Excellent/Very Good | 93 | 98
  2. Good | 2 | 2
  3. Sufficient/Satisfactory | 5 | 0
  4. Unsatisfactory | 0 | 0

7. Secondary Outcome: Fracture of Restorative Material
Description: as for outcome 6
Time Frame: 12 months post-restoration
Population: Six of 51 subjects missed 1-year visit; 1 completed this visit but outside allowed window and was excluded from analysis.
  Scoring categories for this endpoint are:
  1. Excellent/very good: No fractures/cracks
  2. Good: Small hairline cracks
  3. Sufficient/Satisfactory: Two or more or larger hairline cracks and/or material chip fracture not affecting the marginal integrity or approximal contact
  4. Unsatisfactory: Material chip fractures which damage marginal quality or approximal contacts
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 44 | 44
Number analyzed (Restorations) | 44 | 44
percentage of restorations
  1. Excellent/Very Good | 95.4 | 100
  2. Good | 2.3 | 0
  3. Sufficient/Satisfactory | 2.3 | 0
  4. Unsatisfactory | 0 | 0

8. Secondary Outcome: Marginal Adaptation
Description: as for outcome 3
Time Frame: baseline day of restoration
Population: as for outcome 3
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 51 | 51
Number analyzed (Restorations) | 51 | 51
percentage of restorations
  1. Excellent/Very Good | 33 | 37
  2. Good | 67 | 63
  3. Sufficient/Satisfactory | 0 | 0
  4. Unsatisfactory | 0 | 0
  5. Poor | 0 | 0

9. Secondary Outcome: Marginal Adaptation
Description: as for outcome 3
Time Frame: 6 months post-restoration
Population: 10 of 51 subjects missed 6-month visit.
  Scoring categories for this result are:
  1. Excellent/very good: No clinically detectable gap
  2. Good: Marginal integrity deviates from the ideal but could be upgraded to ideal by polishing
  3. Sufficient/satisfactory: Leakage/discoloration is present but limited to the marginal area
  4. Unsatisfactory: Localized major gap that may result in exposure of dentine or base
  5. Poor: Generalized major gap or irregularities; or restoration is loose but in situ
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 41 | 41
Number analyzed (Restorations) | 41 | 41
percentage of restorations
  1. Excellent/Very Good | 22 | 17.1
  2. Good | 76 | 80.5
  3. Sufficient/Satisfactory | 2 | 2.4
  4. Unsatisfactory | 0 | 0
  5. Poor | 0 | 0

10. Secondary Outcome: Marginal Adaptation
Description: as for outcome 3
Time Frame: 12 months post-restoration
Population: 44/51 subjects returned for this visit.
  Scoring categories for this result are:
  1. Excellent/very good: No clinically detectable gap
  2. Good: Marginal integrity deviates from the ideal but could be upgraded to ideal by polishing
  3. Sufficient/satisfactory: Leakage/discoloration is present but limited to the marginal area
  4. Unsatisfactory: Localized major gap that may result in exposure of dentine or base
  5. Poor: Generalized major gap or irregularities; or restoration is loose but in situ
Measure: Number; unit: percentage of restorations
Units Other Than Participants: Restorations
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
Number analyzed (Participants) | 44 | 44
Number analyzed (Restorations) | 44 | 44
percentage of restorations
  1. Excellent/Very Good | 20 | 29.55
  2. Good | 80 | 65.9
  3. Sufficient/Satisfactory | 0 | 4.55
  4. Unsatisfactory | 0 | 0
  5. Poor | 0 | 0

ADVERSE EVENTS:
Time Frame: All device-related and serious adverse events were collected from the time of restoration through the 24-month follow-up visit. Non-serious, non-device related adverse events were collected from the time of restoration through the 6-month follow-up visit.
Arm/Group | Scotchbond Universal Plus Treatment | Scotchbond Universal Comparator
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 8/51 | 8/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scotchbond Universal Plus Treatment (N=51) | Scotchbond Universal Comparator (N=51)
Dental Restoration Failure (General disorders) | 2 (2) | 2 (2) — Complications associated with device not elsewhere classified (NEC). Non-device related adverse event involving a dental restoration or temporary crown on a non-study tooth. NOTE: This event is listed in both groups for a total of 2 events.
Hyperaesthesia teeth (Gastrointestinal disorders) | 2 (2) | 2 (2) — Dental pain and sensation disorders. Non-device related sensitivity of teeth. NOTE: Subjects have two teeth treated with 1 tooth per treatment group. This event is listed in both groups for a total of 2 non-device related events.
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) — Dental and gingival conditions. Dental cavity non-device related. NOTE: Subjects have two teeth treated with 1 tooth per treatment group. This event is listed in both groups but there was 1 non-device related event total.
Gingival Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — Dental and gingival conditions. Gum pain non-device related. NOTE: Subjects have two teeth treated with 1 tooth per treatment group. This event is listed in both groups but there was 1 non-device related event total.
Periodontal Inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1) — Dental and gingival conditions. Periodontal inflammation non-device related. NOTE: Subjects have two teeth treated with 1 tooth per treatment group. This event is listed in both groups but there was 1 non-device related event total.
Tooth Fracture (Gastrointestinal disorders) | 1 (1) | 1 (1) — Dental disorder not elsewhere categorized (NEC) non-device related. NOTE: Subjects have two teeth treated with 1 tooth per treatment group. This event is listed in both groups but there was 1 non-device related event total.
Tooth Infection (Infections and infestations) | 1 (1) | 1 (1) — Dental and Oral soft tissue infections. Non-device related. NOTE: Subjects have two teeth treated with 1 tooth per treatment group. This event is listed in both groups but there was 1 non-device related event total.
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Muscle, tendon and ligament injuries. Ankle sprain non-device related. NOTE: Subjects have two teeth treated with 1 tooth per treatment group. This event is listed in both groups but there was 1 non-device related event total.

LIMITATIONS AND CAVEATS:
Planned randomization of treating pairs of 2 molars or 2 premolars was not always followed. There were 16 subjects who had pairs of 1 molar and 1 premolar treated. These changes were not expected to impact the results of the study and no adjustments to the analysis plan were made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT05248204/Prot_SAP_000.pdf